CLINICAL TRIAL: NCT02016040
Title: Focal Therapy Using High Intensity Focused Ultrasound (ABLATHERM®) for Localised Prostate Cancer
Brief Title: Focal Therapy Using HIFU for Localised Prostate Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr.Franck Bladou, MD. Professor of Oncology and Urology, McGill University, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #12-030
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; HIFU Hemi-ablation; Prostate biopsies
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU hemi-ablation (Active Comparator): Focal Therapy Using High Intensity Focused Ultrasound (Ablatherm)
  Interventions: Procedure: High Intensity Focused Ultrasound

INTERVENTIONS:
Procedure: High Intensity Focused Ultrasound

SUMMARY:
To evaluate the rate of patients without cancer detected by biopsies performed six months after hemi-ablation with high intensity focused ultrasound (HIFU) (Ablatherm ®).

Evaluate the impact of the HIFU treatment on continence, sexuality and quality of life at one year. Evaluate the cost of hemi-ablation HIFU treatment.

A prospective single -centre phase II, single arm, cohort study (therapeutic confirmatory) offering focal therapy using HIFU (Ablatherm ®) to 25 men with histologically proven localised low to intermediate risk prostate cancer (PSA ≤10ng/ml, Gleason score ≤ 7 ,T1c or T2b ). Precise mapping and characterisation of the disease will be established using multi-parametric (mp)-MRI and prostate biopsies. Only the lobe with disease will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 50 years
* Clinical stage T1c (normal digital rectal examination) or T2a (one palpable nodule on digital rectal examination)
* PSA ≤10 ng / mL
* Presence of cancer on biopsies (12 sampling biopsies plus 2-4 targeted biopsies on one side and limited to one or two contiguous areas of prostate: basic and middle or middle and apex).
* Gleason score ≤ 7 (3+4)
* Flowmetry > 12 mL / sec for a voided volume of 125 mL
* PVR <100 mL
* Patient with normal anal and rectal anatomy.
* Patient with a condition corresponding to a classification of ASA 1 or 2.
* Patient signing ICF and agreed for following monitoring

Exclusion Criteria:

* Patient with an ASA score 3.
* Patient in clinical stage T1a, T1b, T2b, T2c or T3.
* Patient with a tumor visible on MRI: Located at a distance less than 5 mm from the midline. Located less than 6 mm from the apex real
* Metastatic lymph node or metastasis discovered by MRI and bone scan.
* Patient previously treated for his prostate cancer by hormone therapy.
* Patient with a distance between the rectal mucosa and prostate capsule over 8 mm thick
* History of inflammatory bowel disease
* Rectal fistula.
* History of pelvic radiotherapy.
* History of bladder cancer.
* History of bladder neck sclerosis or urethral stenosis.
* Patient with an implant located less than 1 cm from the treatment zone (stent, catheter).
* Urogenital infection.
* Latex allergy
* Contraindication to MRI (pacemaker,metal prosthesis ...)
* Patient participated in another clinical study within 30 days.
* Illiterate patients
* Legally incapable patients

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-17 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients without cancer | Six months
  MRI,Biopsy,PSA

SECONDARY OUTCOMES:
Immediate tolerance of hemi-ablation | One year
  Adverse events
Impact of the hemi-ablation HIFU treatment on continence, sexuality and quality of life | One year
  Questionnaires
Cost of hemi-ablation HIFU treatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Franck Bladou, MD, Principal Investigator — Jewish General Hospital,Urology Department
Locations (1):
- Jewish General Hospital,Urology Department, Montreal, Quebec, Canada